CLINICAL TRIAL: NCT00131235
Title: Lungwena Antenatal Intervention Study. A Single-centre Intervention Trial in Rural Malawi, Testing Maternal and Infant Health Effects of Presumptive Intermittent Treatment of Pregnant Women With Sulfadoxine-pyrimethamine and Azithromycin
Brief Title: Gestational Sulfadoxine-pyrimethamine and Azithromycin Treatment to Prevent Preterm Birth
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Academy of Finland (Other); Foundation for Paediatric Research, Finland (Other)
Responsible Party: Principal Investigator, Per Ashorn, Professor of Pediatrics, Tampere University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SA-179787-1
Record Dates: First submitted 2005-08-16; First posted 2005-08-17 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Malaria; Sexually Transmitted Diseases; Preterm Birth; Pregnancy
Keywords: Malaria; STI; Pregnancy; Prevention; Preterm birth; Low birth weight; Sub-Saharan Africa
MeSH Terms: conditions — Malaria; Sexually Transmitted Diseases; Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Placebo Comparator): Standard antenatal care as described in intervention
  Interventions: Drug: Sulfadoxine-pyrimethamine treatment twice during pregnancy
- Monthly SP (Experimental): Standard antenatal care + monthly intermittent presumptive treatment of malaria with sulfadoxine pyrimethamine, as described in intervention
  Interventions: Drug: Sulfadoxine-pyrimethamine at 4-week intervals
- AZI-SP (Experimental): Standard antenatal care + monthly intermittent presumptive treatment of malaria with sulfadoxine pyrimethamine + two presumptive treatments of sexually transmitted infections and malaria with azithromycin, as described in intervention
  Interventions: Drug: Sulfadoxine-pyrimethamine every 4 weeks + azithromycin twice

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine treatment twice during pregnancy — Sulfadoxine-pyrimethamine, 3 tablets (each containing 500mg of sulfadoxine and 25mg of pyrimethamine), taken once at antenatal care enrolment (14.0-25.9 gestation weeks) and another time between 28.0 and 33.9 gestation weeks.
  2 placebo tablets for azithromycin taken at the same time points.
  Other Names: Control
  Arms: Control
Drug: Sulfadoxine-pyrimethamine at 4-week intervals — Sulfadoxine-pyrimethamine, 3 tablets (each containing 500mg of sulfadoxine and 25mg of pyrimethamine), taken once at antenatal care enrolment (14.0-25.9 gestation weeks) and then at 4 week intervals until 37.0 gestation weeks.
  2 placebo tablets for azithromycin taken once at antenatal care enrolment (14.0-25.9 gestation weeks) and another time between 28.0 and 33.9 gestation weeks.
  Other Names: Monthly SP
  Arms: Monthly SP
Drug: Sulfadoxine-pyrimethamine every 4 weeks + azithromycin twice — Sulfadoxine-pyrimethamine, 3 tablets (each containing 500mg of sulfadoxine and 25mg of pyrimethamine), taken once at antenatal care enrolment (14.0-25.9 gestation weeks) and then at 4 week intervals until 37.0 gestation weeks.
  2 azithromycin tablets (each 500 mg) taken once at antenatal care enrolment (14.0-25.9 gestation weeks) and another time between 28.0 and 33.9 gestation weeks.
  Other Names: Azi-SP
  Arms: AZI-SP

SUMMARY:
The purpose of this study is to examine whether treatment of pregnant Malawian women with repeated doses of sulfadoxine-pyrimethamine and azithromycin antibiotics will prevent preterm deliveries and result in other health benefits both for the mother and the foetus/newborn.

DETAILED DESCRIPTION:
Maternal anaemia, preterm deliveries and low birth weight are common in Sub-Saharan Africa and contribute significantly to the ill-health of pregnant women and infants. The present study is based on the assumption that these adverse outcomes can be prevented by improved antimicrobial management of malaria and sexually transmitted infections (STI) among pregnant women. To test the hypothesis, a randomised clinical trial following Good Clinical Practice (GCP) is being carried out in Malawi, South-Eastern Africa.

A total of 1320 consenting women who present at a rural antenatal clinic after 14 but before 26 completed gestation weeks will be enrolled. One third of the women will receive antenatal care according to national recommendations, including regular visits to health centre, screening for pregnancy complications, haematinic and vitamin A supplementation and two doses of presumptive malaria treatment with sulfadoxine-pyrimethamine. Another third will receive otherwise the same care, but sulfadoxine-pyrimethamine treatment is given at monthly intervals. The final third receives standard antenatal care, sulfadoxine-pyrimethamine treatment at monthly intervals and two doses of presumptive STI treatment with azithromycin. Women are monitored throughout pregnancy and delivery and newborn growth will be followed up for five years.

The primary outcome measure is proportion of preterm births in the three study groups. Secondary maternal outcomes include anaemia and malaria parasitaemia during pregnancy, at delivery and at 1, 3, and 6 months after delivery, gestational weight gain and morbidity and STI prevalence after delivery. Secondary child outcomes consist of proportion of babies with low birth weight, mean birth weight, growth in infancy and childhood, incidence of malnutrition in infancy and childhood, and mortality. Additionally, information is collected on the development of malaria-specific humoral immunity in pregnancy and participant experiences from the study. Participant safety is systematically monitored throughout the intervention.

There have been two edits two the trial protocol, since the original approval. In the first one, there was an amendment to follow child growth and mortality until and child development at 5 years of age, with visits at 1, 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 48, and 60 months. In the second amendment, there was an addition to monitor child antropometrics, physical, mental, and social health at and mortality by 10-12 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age >= 15 years
* Ultrasound confirmed pregnancy
* Quickening
* Foetal age 14-26 gestation weeks
* Maternal availability for follow-up during the entire study period

Exclusion Criteria:

* Known maternal tuberculosis, diabetes, kidney disease or liver disease
* Any severe acute illness warranting hospital referral at enrollment visit
* Mental disorder that may affect comprehension of the study or success of follow-up
* Twin pregnancy
* Pregnancy complications evident at enrollment visit (moderate to severe oedema, blood hemoglobin [Hb] concentration < 50 g/l, systolic blood pressure [BP] > 160 mmHg or diastolic BP > 100 mmHg)
* Prior receipt of azithromycin during this pregnancy
* Receipt of sulfadoxine and pyrimethamine within 28 days of enrollment
* Known allergy to drugs containing sulfonamides, macrolides or pyrimethamine
* History of anaphylaxis
* History of any serious allergic reaction to any substance, requiring emergency medical care
* Concurrent participation in any other clinical trial

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1320 (Actual)
Dates: Start 2003-12; Primary Completion 2007-06 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of preterm births | once, after delivery
  Proportion of babies who are born before 37 completed gestation weeks
Number of serious adverse events | Cumulative during pregnancy and neonatal period
  Death, life-threatening event, hospitalization, congenital anomaly, or any othe condition consedered an SAE by a study physician

SECONDARY OUTCOMES:
Percentage of low birth weight babies | Once, after delivery
  Birth weight < 2500 g
Mean birth weight | Once, after delivery
  Measured in grams
Mean duration of gestation | Once, after delivery
  Measured in gestation weeks, expressed to one deciman,
Percentage of low head circumference at birth | Once, after delivery
  Below 2 standard deviations of the mean of international reference population
Incidence of moderate underweight during infancy or childhood | Cumulative during infancy and childhood
  weight for age Z-score < -2
Perinatal mortality | Cumulative until 7 days of post-natal life
  Stillbirths after 22 gestation weeks or within first 7 days of life / 1000 live births
Neonatal mortality | Cumulative until 28 days of post-natal life
  Deaths within first 28 days of life / 1000 live births
Infant mortality | Cumulative until 365 days of post-natal life
  Deaths within first 265 days of life / 1000 live births
Mean maternal blood haemoglobin concentration at each antenatal visit and at 1, 3, and 6 months after delivery | Several antenatal and postnatal visits
  Measured with hemocue meter, expressed as grams / liter
Percentage of women with mild, moderate or severe anaemia at every antenatal visit and at 1, 3, and 6 months after delivery | Several antenatal and postnatal visits
  Cut-offs for mild, moderate and severa anaemia 110 g / l - 80 g / l - 50 g / l
Percentage of women with peripheral blood malaria parasitaemia at 32 gestational weeks and at delivery | At enrolment, every 4 weeks thereafter and at delivery
  Measured with microscopy from fresh blood slides and with real-time PCR from dried blood spots
Maternal weight gain during pregnancy | Cumulative during pregnancy
  grams / gestation week
Mean number of maternal illness days during pregnancy | Cumulative during pregnancy
  Self reported illness symptoms
Prevalence of maternal chlamydia trachomatis, neisseria gonorrhoea, and vaginal trichomoniasis infection at 4 weeks after delivery | At 4 weeks after delivery
  Chlamydia and gonorhoea measured from urine samples with a PCR, vaginal trichomoniasis measures with a wet microscopy
Attained lenght / height | 1, 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 48, 60 months and 10-12 years of age
  Measured as length until 2 years of age, then height; expressed in cm (one decimal) and as length / heigh for age Z-score
Attained weight | 1, 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 48, 60 months and 10-12 years of age
  Expressed in kg with two decimals and as weight for age Z-score
Nutritional status | 1, 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 48, 60 months and 10-12 years of age
  Mid-upper arm circumference, in mm (no decimals)
Attained head circumference | 1, 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 48, 60 months and 10-12 years of age
  Head circumference, in mm, no decimals
Childhood mortality, % of subjects who have died by the 10-12 year follow-up visit | Cumulative incidence by 10-12 years of age
  Deaths, information obtained from parents or other adults who have lived in the same household with the child
Motor development, Griffiths test, sub-score | 5 years of age
  Summary score from questions in the gross motor and fine motor domain questions
Social development, Griffiths test, sub-score | 5 years of age
  Summary score from questions in the social development domain questions
Cognitive development, Raven's colour matrix, score | 10-12 years of age
  Summary score from 36 questions in the Raven's colour matrix test
Reaction time, milliseconds | 10-12 years of age
  This will be tested with an eye-tracking device (Tobii). Participants are asked to look from the fixation point to different directions or fixate the gaze at one point. We will measure the horizontal eye-movements (saccades) and calculate the reaction times, scoring the task correct/incorrect (direction).
  This eye-tracking system is based on a Pupil Centre Corneal Reflection (PCCR) technique, in which near infrared illumination is reflected on the cornea relative to the center of the pupil. The eye-tracking cameras capture the light reflections and create a 3D model of the eye and head-position to track the participant's point of gaze at high temporal and spatial accuracy (60 Hz/0.4°). The results will be stored automatically into a data base.
Systolic blood pressure, mmHg | 10-12 years of age
  Will use oscillometric Mobil o Graph blood pressure monitoring system (accuracy +/- 3 mmHg), when the child is first sitting, then standing and last lying down.
Diastolic blood pressure, mmHg | 10-12 years of age
  Will use oscillometric Mobil o Graph blood pressure monitoring system (accuracy +/- 3 mmHg), when the child is first sitting, then standing and last lying down.
Central blood pressure, mmHg | 10-12 years of age
  Will use oscillometric Mobil o Graph blood pressure monitoring system (accuracy +/- 3 mmHg), when the child is first sitting, then standing and last lying down.
Pulse rate, beats / minutes | 10-12 years of age
  Will use oscillometric Mobil o Graph blood pressure monitoring system. We will measure pulse rate / minutes, when the child is first sitting, then standing and last lying down.
Vascular resistance, mmHg·min/l | 10-12 years of age
  Will use oscillometric Mobil o Graph blood pressure monitoring system. We will measure vascular resistance, when the child is first sitting, then standing and last lying down.
Lean body mass, expressed in kg, with one decimal | 10-12 years of age
  Body composition measured with 8-polar biompedance method (Seca® mBCA 515 Medical Body Composition Analyser), validated with Deuterium Dilution Technique with Analysis of Saliva Samples by Fourier Transform Infrared Spectrometry (FTIR)
Fat mass, expressed in kg, with one decimal | 10-12 years of age
  Body composition measured with 8-polar biompedance method (Seca® mBCA 515 Medical Body Composition Analyser), validated with Deuterium Dilution Technique with Analysis of Saliva Samples by Fourier Transform Infrared Spectrometry (FTIR)
Fat percentage, expressed proportion of body weight (per cent, with one decimal) | 10-12 years of age
  Body composition measured with 8-polar biompedance method (Seca® mBCA 515 Medical Body Composition Analyser), validated with Deuterium Dilution Technique with Analysis of Saliva Samples by Fourier Transform Infrared Spectrometry (FTIR)
Self-rated well-being, score | 10-12 years of age
  Self-reported well-being will be measured with 11 question panel with rating from 1-5 expressed as smileys. The questions consider about "how happy you are about the things you own, school, house you live, food, clothes, other pupils, friends, the family, safety feeling, the way you look, with yourself". Score for self-reported well-being will be calculated as a sum of ratings for each item divided by the number of items with non-missing data. There are two items related to the child's school and they are not applicable if the child does not go to school. The minimum score for self-reported well-being is 1 and the maximum is 5, and the score will be expressed with one decimal.

CONTACTS AND LOCATIONS:
Overall Officials: Per Ashorn, MD, PhD, Study Director — Tampere University, Faculty of Medicine and Health Technology; Kenneth M Maleta, MBBS, PhD, Principal Investigator — Kamuzu University of Health Sciences
Locations (1):
- College of Medicine, University of Malawi, Mangochi, Mangochi District, Malawi

REFERENCES:
- [Background] Kayentao K, Garner P, van Eijk AM, Naidoo I, Roper C, Mulokozi A, MacArthur JR, Luntamo M, Ashorn P, Doumbo OK, ter Kuile FO. Intermittent preventive therapy for malaria during pregnancy using 2 vs 3 or more doses of sulfadoxine-pyrimethamine and risk of low birth weight in Africa: systematic review and meta-analysis. JAMA. 2013 Feb 13;309(6):594-604. doi: 10.1001/jama.2012.216231. PMID 23403684
- [Background] Hallamaa L, Cheung YB, Maleta K, Luntamo M, Ashorn U, Gladstone M, Kulmala T, Mangani C, Ashorn P. Child Health Outcomes After Presumptive Infection Treatment in Pregnant Women: A Randomized Trial. Pediatrics. 2018 Mar;141(3):e20172459. doi: 10.1542/peds.2017-2459. PMID 29472491
- [Result] Luntamo M, Kulmala T, Mbewe B, Cheung YB, Maleta K, Ashorn P. Effect of repeated treatment of pregnant women with sulfadoxine-pyrimethamine and azithromycin on preterm delivery in Malawi: a randomized controlled trial. Am J Trop Med Hyg. 2010 Dec;83(6):1212-20. doi: 10.4269/ajtmh.2010.10-0264. PMID 21118924
- [Result] Rantala AM, Taylor SM, Trottman PA, Luntamo M, Mbewe B, Maleta K, Kulmala T, Ashorn P, Meshnick SR. Comparison of real-time PCR and microscopy for malaria parasite detection in Malawian pregnant women. Malar J. 2010 Oct 6;9:269. doi: 10.1186/1475-2875-9-269. PMID 20925928
- [Result] Aitken EH, Mbewe B, Luntamo M, Kulmala T, Beeson JG, Ashorn P, Rogerson SJ. Antibody to P. falciparum in pregnancy varies with intermittent preventive treatment regime and bed net use. PLoS One. 2012;7(1):e29874. doi: 10.1371/journal.pone.0029874. Epub 2012 Jan 27. PMID 22299027
- [Result] Aitken EH, Mbewe B, Luntamo M, Maleta K, Kulmala T, Friso MJ, Fowkes FJ, Beeson JG, Ashorn P, Rogerson SJ. Antibodies to chondroitin sulfate A-binding infected erythrocytes: dynamics and protection during pregnancy in women receiving intermittent preventive treatment. J Infect Dis. 2010 May 1;201(9):1316-25. doi: 10.1086/651578. PMID 20350189
- [Result] Luntamo M, Kulmala T, Cheung YB, Maleta K, Ashorn P. The effect of antenatal monthly sulphadoxine-pyrimethamine, alone or with azithromycin, on foetal and neonatal growth faltering in Malawi: a randomised controlled trial. Trop Med Int Health. 2013 Apr;18(4):386-97. doi: 10.1111/tmi.12074. Epub 2013 Feb 22. PMID 23432801
- [Result] Xu J, Luntamo M, Kulmala T, Ashorn P, Cheung YB. A longitudinal study of weight gain in pregnancy in Malawi: unconditional and conditional standards. Am J Clin Nutr. 2014 Feb;99(2):296-301. doi: 10.3945/ajcn.113.074120. Epub 2013 Nov 13. PMID 24225354
- [Result] Lin JT, Mbewe B, Taylor SM, Luntamo M, Meshnick SR, Ashorn P. Increased prevalence of dhfr and dhps mutants at delivery in Malawian pregnant women receiving intermittent preventive treatment for malaria. Trop Med Int Health. 2013 Feb;18(2):175-8. doi: 10.1111/tmi.12028. Epub 2012 Nov 30. PMID 23198734
- [Derived] Pons-Duran C, Wassenaar MJ, Yovo KE, Marin-Carballo C, Briand V, Gonzalez R. Intermittent preventive treatment regimens for malaria in HIV-positive pregnant women. Cochrane Database Syst Rev. 2024 Sep 26;9(9):CD006689. doi: 10.1002/14651858.CD006689.pub3. PMID 39324693
- [Derived] Videman K, Hallamaa L, Heimonen O, Mangani C, Luntamo M, Maleta K, Ashorn P, Ashorn U. Child growth and neurodevelopment after maternal antenatal antibiotic treatment. Arch Dis Child. 2022 Apr;107(4):323-328. doi: 10.1136/archdischild-2021-322043. Epub 2021 Sep 3. PMID 34479861
- [Derived] Luntamo M, Rantala AM, Meshnick SR, Cheung YB, Kulmala T, Maleta K, Ashorn P. The effect of monthly sulfadoxine-pyrimethamine, alone or with azithromycin, on PCR-diagnosed malaria at delivery: a randomized controlled trial. PLoS One. 2012;7(7):e41123. doi: 10.1371/journal.pone.0041123. Epub 2012 Jul 19. PMID 22829919
- See also: College of Medicine home page — http://www.medcol.mw/